CLINICAL TRIAL: NCT00407277
Title: Neural Inhibition as a Mechanism of Nicotine Dependence Among Persons With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Psychiatric Research Foundation (Other)
Responsible Party: Dr. Jeff Daskalakis, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 63/2005
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Smoking; Nicotine Dependence; Schizophrenia; Schizophreniform Disorders; Schizoaffective Disorder; Psychosis
Keywords: nicotine dependence; smoking; nicotine patch; double-blind; randomized; placebo; psychosis; schizophrenia; schizophreniform; schizoaffective disorder
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Schizophrenia; Psychotic Disorders | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1A (Experimental)
  Interventions: Drug: Nicotine patch
- 1B (Placebo Comparator)
  Interventions: Other: placebo
- 2A (Experimental)
  Interventions: Behavioral: smoking cessation group therapy

INTERVENTIONS:
Drug: Nicotine patch — 21 mg of nicotine via a dermal patch
  Arms: 1A
Other: placebo — placebo via a dermal patch
  Arms: 1B
Behavioral: smoking cessation group therapy — a 9-week group based on the "Freedom From Smoking" program designed by the American Lung Association. The treatment was manualized and modified to meet the functional and cognitive capabilities of patients with psychotic disorders
  Arms: 2A

SUMMARY:
Cigarette smoking decreases life expectancy, causes devastating health complications, and costs society billions of dollars each year. These untoward consequences are especially pronounced among persons with schizophrenia (SCZ) because approximately 80% to 95% of this group smokes cigarettes. These high prevalence rates underscore the need for research investigating the determinants of smoking in patients with SCZ. Several researchers have observed that nicotine improves specific symptoms of SCZ including negative symptoms, negative affect, and cognitive deficits. This has led to the hypothesis that patients with SCZ smoke in an attempt to self-medicate. However, the mechanism(s) by which nicotine has its positive effect on symptoms remains unclear. The current proposal posits that neural inhibition (NI) is a physiological mechanism of this effect, while variation in the alpha-7-nicotinic receptor subunit gene (CHRNA7) represents the genetic underpinnings of these processes. The proposed study will assess NI and symptom improvement after acute administration of nicotine to both smokers and nonsmokers with SCZ. In addition, NI and CHRNA7 variation will be tested as predictors of patients' ability to reduce/quit smoking following smoking treatment. These data may lead to the development of new pharmacological strategies for treating the symptoms of SCZ and new methods for assisting these patients to quit smoking.

DETAILED DESCRIPTION:
The prevalence of smoking is unusually high among patients with SCZ. In light of the negative health, economic, and social consequences of smoking, treatment efforts in this area are imperative. Such efforts rest, in part, on an improved understanding of the underlying causes of smoking within this unique population. For example, several lines of research have indicated that smoking improves specific SCZ-related symptoms (i.e., negative psychotic symptoms, negative affect, cognitive deficits) and that patients may smoke to self-medicate with nicotine. However, the mechanism(s) underlying this effect are unknown. The current proposal posits that improved NI may be one such mechanism. More specifically, NI is conceived as a mediator of the relationship between smoking and symptom improvement. Also, given its proposed mechanistic nature, we believe that nicotine-related changes in NI may predict quit/reduction and/or relapse rates following a smoking cessation program. Additionally, variants of CHRNA7 likely represent the genetic underpinnings of decreased NI, vulnerability to smoking, and smoking treatment resistance among patients with SCZ. These hypotheses are supported by previous experiments that suggest: (1) patients with SCZ have decreased NI (Adler et al., 1998); (2) nicotine administration (via its effects on the alpha-7-nicotinic receptor, which, in turn activates GABAergic interneurons) enhances NI in these patients (Adler et al., 1998); (3) genetic variation in the alpha-7-nicotinic receptor increases risk for smoking among patients with SCZ (Leonard et al., 1996); and, (4) higher levels of NI are associated with fewer negative symptoms, less negative affect, and better cognition (Yee et al., 1998). However, these studies have been hampered by several methodological and conceptual shortcomings including small sample sizes, the presence of confounding variables (e.g., the effects of nicotine withdrawal), and limited testing of relevant symptom domains. Furthermore, previous studies have examined only isolated aspects of the proposed model, leaving many of the central relationships between variables untested and speculative. The current proposal seeks to rectify these methodological issues within the context of a multidisciplinary scientific team. Globally, its objectives are twofold. First, to replicate and extend previous findings that nicotine causes symptom attenuation. Second to investigate the underlying neurophysiological and genetic mechanisms of these effects. The specific objectives and hypotheses addressed in this study are as follows:

1. To acutely administer nicotine versus placebo to smokers with SCZ following transient abstinence from cigarettes, in order to investigate the effect of nicotine on the SCZ symptoms. This objective extends previous research by employing an adequately large sample and simultaneously testing several relevant domains of symptom improvement. Hypothesis: Significantly greater improvements across the domains of negative symptoms, negative affect, and cognitive deficits will be evident among those patients receiving nicotine versus placebo.
2. To acutely administer nicotine versus placebo to nonsmokers with SCZ in order to investigate the effects of nicotine on the symptoms of SCZ, independent of withdrawal. This objective allows for the methodological disambiguation of the direct neural effects of nicotine from the effects of termination of withdrawal symptoms. Additionally, this will provide seminal data regarding the acute treatment benefits of nicotine as a therapeutic agent, delivered without the health risks associated with smoking. Hypothesis: Significantly greater improvements across all symptoms domains will be evident among those patients receiving nicotine versus placebo.
3. To ascertain (using statistical techniques outlined by Kenny and others) (Baron & Kenny, 1986; Judd &Kenny, 1981) whether the relationship between acute nicotine administration and symptom reductions is mediated by increased NI (as measured via ERP and TMS paradigms). Hypothesis: NI will meet the statistical criteria for mediating the relationship between nicotine administration and symptom reductions.
4. To ascertain whether nicotine-related changes in NI predict patients' ability to reduce smoking, the amount of nicotine replacement therapy (NRT) required, and rates of quitting and smoking relapse following completion of a smoking cessation program. Hypothesis: NI will operate as a significant and unique predictor of the amount of smoking reduction and NRT use, as well as quit and relapse rates, over and above conventional predictors of smoking reduction from the general population (i.e., age, marital status, coping resources, socioeconomic status, smoking related health problems, the number of cigarettes smoked per day, concomitant alcohol and coffee consumption, treatment compliance, and stage of change) (Matheny & Weatherman, 1998; Ockene et al., 2000; Oritz et al., 2003).
5. To investigate whether polymorphisms in CHRNA7 are associated with the magnitude of NI deficits, symptom reductions following acute nicotine administration, rates of smoking among patients with SCZ, and/or quit/reduction or relapse rates following smoking cessation treatment. Hypothesis: Significant genetic association will be demonstrated between CHRNA7 polymorphisms and each of the above-listed clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and competent to consent
* Have a diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder as confirmed by the Structured Clinical Interview for the DSM-IV (SCID-IV)
* Between the ages of 18 and 60

Exclusion Criteria:

* Have a DSM-IV history of substance abuse or dependence (other than caffeine or nicotine) in the last 6 months
* Have a self-reported concomitant major medical or neurologic illness
* Pregnant
* Currently prescribed medications known to deleteriously affect cognition (e.g., benzodiazepines, tricyclic anti-depressants, anticholinergics, MAO inhibitors, GABA-B agonists)
* Currently taking clozapine (due to its documented effect on both NI and smoking
* Report suffering from conditions that may be aggravated by acute nicotine administration (e.g., arrhythmias, recent myocardial infarction)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
neural inhibition via EEG and TMS | intermittent

SECONDARY OUTCOMES:
Self reported tobacco use | intermittent
Polymorphic markers in the CHRNA7 gene and promoter region | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Daskalakis, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Addington J, el-Guebaly N. Group treatment for substance abuse in schizophrenia. Can J Psychiatry. 1998 Oct;43(8):843-5. doi: 10.1177/070674379804300810. PMID 9806092
- [Background] Addington J, el-Guebaly N, Campbell W, Hodgins DC, Addington D. Smoking cessation treatment for patients with schizophrenia. Am J Psychiatry. 1998 Jul;155(7):974-6. doi: 10.1176/ajp.155.7.974. PMID 9659869
- [Background] Addington D, Addington J, Maticka-Tyndale E. Assessing depression in schizophrenia: the Calgary Depression Scale. Br J Psychiatry Suppl. 1993 Dec;(22):39-44. PMID 8110442
- [Background] Adler LE, Olincy A, Waldo M, Harris JG, Griffith J, Stevens K, Flach K, Nagamoto H, Bickford P, Leonard S, Freedman R. Schizophrenia, sensory gating, and nicotinic receptors. Schizophr Bull. 1998;24(2):189-202. doi: 10.1093/oxfordjournals.schbul.a033320. PMID 9613620
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Bohadana A, Nilsson F, Rasmussen T, Martinet Y. Nicotine inhaler and nicotine patch as a combination therapy for smoking cessation: a randomized, double-blind, placebo-controlled trial. Arch Intern Med. 2000 Nov 13;160(20):3128-34. doi: 10.1001/archinte.160.20.3128. PMID 11074742
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research